CLINICAL TRIAL: NCT00692796
Title: Pulmonary Rehabilitation for Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Mordecai Palliative Care Research Fund (Unknown)
Responsible Party: Jeff Swigris, DO, MS, National Jewish Medical and Research Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: NJMRC HS 1603 substudy
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary fibrosis; Pulmonary rehabilitation; Dyspnea; Quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pulmonary rehabilitation is a multi-disciplinary program that includes exercise training, disease education, psychosocial education (e.g., stress management, coping with chronic illness) and nutrition education.

SUMMARY:
The purpose of this study is to determine the effects of Pulmonary Rehabilitation (PR) on shortness of breath, exercise capacity, symptom control, mental health, cognitive function, and quality of life in patients with Idiopathic Pulmonary Fibrosis (IPF). Pulmonary rehabilitation has already been shown to benefit patients with other chronic respiratory diseases, such as chronic obstructive pulmonary disease (COPD). We believe that pulmonary rehabilitation will benefit patients with IPF as well.

DETAILED DESCRIPTION:
The goals of this project are to assess the effect of PR on a number of important outcomes in patients with IPF. Once enrolled in the study, subjects will complete a battery of questionnaires and tests that assess symptoms, quality of life, cognition, and mental health, and then subjects will complete a six week outpatient PR program (at National Jewish Medical and Research Center or other PR programs). Subjects will complete the same battery of questionnaires and tests immediately after completion of the PR program and again six months later.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Diagnosis of IPF according to American Thoracic Society criteria

Exclusion criteria:

* Patients who have completed a PR program within the last two years
* Patients with unstable medical conditions that would make PR unsafe

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 6 weeks and again at 6 months

SECONDARY OUTCOMES:
Cognition | 6 weeks and again at 6 months
Quality of life | 6 weeks and again at 6 months
Fatigue | 6 weeks and again at 6 months
Anxiety | 6 weeks and again at 6 months
Depression | 6 weeks and again at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Swigris, DO, MS, Principal Investigator — National Jewish Medical and Research Center (Jeffrey J. Swigris, DO, MS; Assistant Professor of Medicine)
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Swigris JJ, Fairclough DL, Morrison M, Make B, Kozora E, Brown KK, Wamboldt FS. Benefits of pulmonary rehabilitation in idiopathic pulmonary fibrosis. Respir Care. 2011 Jun;56(6):783-9. doi: 10.4187/respcare.00939. Epub 2011 Feb 11. PMID 21333082